CLINICAL TRIAL: NCT06866652
Title: Evaluating Dyspnea in Autoimmune Myasthenia Gravis "Why am I Short of Breath?"
Acronym: MyaRESP
Status: Not yet recruiting | Type: Observational
Sponsor: Institut de Myologie, France (Other)
Collaborators: APHP (Other)
Responsible Party: Sponsor
Other Study IDs: MyaRESP
Record Dates: First submitted 2025-02-20; First posted 2025-03-10 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Myasthenia Gravis; Dyspnea
Keywords: dyspnea; breathlessness; respiratory
MeSH Terms: conditions — Myasthenia Gravis; Dyspnea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Individuals with MG (IwMG) experience shortness of breath that may be activity-related, occur at rest and even happen during sleep. Dyspnea is a complex, multidimensional and multifactorial symptom involving sensory perception, cognition and emotion. Identifying the cause(s) of dyspnea in MG may assist in finding therapeutic strategies, reducing discomfort, improving QoL and potentially limiting respiratory deterioration and incidence of MG crisis.

DETAILED DESCRIPTION:
MYaResp is a prospective observational, cross-sectional study to evaluate dyspnea in adults with autoimmune myasthenia gravis.

Study aims include to:

* Describe the characteristics of dyspnea in IwMG
* Understand contributing factors and factors associated with dyspnea in IwMG including the relationship between patient-reported dyspnea, disease severity and functional limitations.
* Determine the most effective tests to identify the causes and contributing factors of dyspnea

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* Confirmed diagnosis of autoimmune MG
* Shortness of breath in daily life: score 1 or 2 on the respiration item on the MG- activities of daily living score
* Signed consent form
* Affiliated to or beneficiary of a social security scheme

Exclusion Criteria:

* Known Pregnancy
* Known respiratory disorder (other than MG)
* Recent (within past 4 weeks) respiratory infection
* Current MG crisis or exacerbation (necessitating increase in MG medication &/or hospital admission)
* No dyspnea - score 0 or 3 on the respiration item on the MG- activities of daily living score
* Severe cognitive impairment/guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Age ≥18 Confirmed diagnosis of autoimmune MG Shortness of breath in daily life: score 1 or 2 on the respiration item on the MG- activities of daily living score
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Dyspnea questionnaires | baseline
  Dyspnea-12

SECONDARY OUTCOMES:
cardiopulmonary exercise test | baseline
  cycle ergometer
Polysomnography | baseline
  evaluation of sleep disordered breathing
Functional measures | baseline
  6 minute walk test
Quality of life questionnaires | baseline
  Revised version of the myasthenia gravis quality of life questionnaire (Burns, French validation Birnbaum)
Anxiety and depression | baseline
  Hospital Anxiety and Depression Scale

OTHER OUTCOMES:
impact of myasthenia in daily living | baseline
  impact of myasthenia in daily living score
Respiratory pressures | baseline
  inspiratory and expiratory pressures

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Myology, Paris, France

IPD SHARING:
Plan to Share IPD: No